CLINICAL TRIAL: NCT00525772
Title: Effect of Ciclesonide on Exercise Induced Bronchoconstriction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Kolding Sygehus (Other); Takeda (Industry)
Responsible Party: Paul O'Byrne, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BY/M1-121; OBCIEX
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Last update posted 2009-10-21 (Estimated); Status verified 2009-10

CONDITIONS: Asthma
Keywords: asthma; exercise induced bronchoconstriction; sputum eosinophils
MeSH Terms: conditions — Asthma | interventions — ciclesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): ciclesonide 50 and 200ug
  Interventions: Drug: ciclesonide
- 2 (Active Comparator): ciclesonide 100ug and 400ug
  Interventions: Drug: ciclesonide

INTERVENTIONS:
Drug: ciclesonide — low dose- 50ug and 200ug
  Other Names: ciclesonide (Alvesco)
  Arms: 1
Drug: ciclesonide — high dose- 100ug and 400ug
  Other Names: ciclesonide (Alvesco)
  Arms: 2

SUMMARY:
The purpose of this study is to study the effects of once daily inhaled ciclesonide at varying doses on exercise provoked asthma symptoms, fall in lung function after exercise and sputum characteristics.

DETAILED DESCRIPTION:
To study the effects of 4 doses of ciclesonide on exercise-induced bronchoconstriction, bronchial responsiveness to mannitol, sputum parameters and other parameters of asthma control in asthmatic patients. The primary aim was to evaluate exercise-induced bronchoconstriction as a method of determining the dose and time responses of inhaled corticosteroid therapy. The secondary aims were to evaluate the dose and time responses of sputum parameters and responsiveness to mannitol to inhaled corticosteroid therapy. Furthermore to explore the relationship(s) between exercise induced bronchoconstriction, sputum parameters and mannitol responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* stable asthma not on maintenance asthma medications
* exercise induced bronchoconstriction on dry air exercise challenge.

Exclusion Criteria:

* other significant co-morbidity or treatments that might interfere with the conduct or results of the study
* fail to return to baseline after a maximum washout period of 8 weeks
* unable to perform the procedures of the study

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2001-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
change in maximum fall in FEV1 induced by dry air exercise challenge after treatment compared to the respective pretreatment value | at 1 week of treatment

SECONDARY OUTCOMES:
Changes in sputum cell counts,bronchial responsiveness to mannitol and other clinical parameters of asthma control after treatment compared to respective pre-treatment value. | after 1, 2, 3, weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paul O'Byrne, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Subbarao P, Duong M, Adelroth E, Otis J, Obminski G, Inman M, Pedersen S, O'byrne PM. Effect of ciclesonide dose and duration of therapy on exercise-induced bronchoconstriction in patients with asthma. J Allergy Clin Immunol. 2006 May;117(5):1008-13. doi: 10.1016/j.jaci.2005.11.048. PMID 16675326
- [Derived] Duong M, Subbarao P, Adelroth E, Obminski G, Strinich T, Inman M, Pedersen S, O'Byrne PM. Sputum eosinophils and the response of exercise-induced bronchoconstriction to corticosteroid in asthma. Chest. 2008 Feb;133(2):404-11. doi: 10.1378/chest.07-2048. Epub 2007 Dec 10. PMID 18071011